CLINICAL TRIAL: NCT07026747
Title: The Effects of Core Stabilization Exercises on Functional and Emotional Status in Traumatic Hand Injuries
Brief Title: Effects of Core Stabilization on Hand Trauma Outcomes
Acronym: TH-CORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstinyeUni-B.UYANIK.001
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Hand Injuries
Keywords: hand injuries; core stabilization exercise; function; emotion
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial includes three parallel groups designed to compare the effects of: standard hand rehabilitation alone, standard hand rehabilitation combined with supervised core stabilization exercises, and standard hand rehabilitation combined with unsupervised core stabilization exercises delivered via pre-recorded video.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Hand Rehabilitation Only (Active Comparator): This control group will receive the standard hand rehabilitation program.
  Interventions: Behavioral: Standard Hand Rehabilitation Only
- Supervised Core Stabilization + Standard Hand Rehabilitation (Experimental): This group will perform core exercises supervised by a physiotherapist in addition to the standard hand rehabilitation program.
  Interventions: Behavioral: Supervised Core Stabilization + Standard Hand Rehabilitation
- Unsupervised Core Stabilization + Standard Hand Rehabilitation (Experimental): This group will perform the same core exercises as the second group by watching videos in the same clinical setting.
  Interventions: Behavioral: Unsupervised Core Stabilization + Standard Hand Rehabilitation

INTERVENTIONS:
Behavioral: Standard Hand Rehabilitation Only — Standard Hand Rehabilitation Program will be delivered over a total duration of six weeks. During the first three weeks, the program will be administered five days per week, and during the following three weeks, it will be performed three days per week. The rehabilitation program will include scar tissue massage, passive and active range of motion exercises for the fingers and wrist, sensory re-education, and edema control using retrograde massage and Coban wrapping. Joint mobilization techniques will be applied to the finger and wrist joints, along with tendon gliding and tendon blocking exercises. Strengthening and stretching exercises targeting the hand and wrist muscles will be progressively introduced throughout the program. Functional training and moderate-level activities will be included as tolerated, particularly in the later stages of the program. The intervention will be structured to gradually increase in intensity and complexity across three phases, each lasting two weeks.
  Arms: Standard Hand Rehabilitation Only
Behavioral: Supervised Core Stabilization + Standard Hand Rehabilitation — The second group will receive the same six-week Standard Hand Rehabilitation Program as the control group (5 days per week for the first 3 weeks, and 3 days per week for the last 3 weeks). In addition, participants will perform a Supervised Core Stabilization Exercise Program three times per week for six weeks under a physiotherapist's supervision.The exercises will focus on activating the transversus abdominis and coordinating breathing to improve core stability.Each session will include a warm-up, main core exercises, and a cool-down.In weeks 0-2, the program will include diaphragmatic breathing, transversus abdominis activation, curl-ups, and bridging. In weeks 2-4, it will progress to cross arm-leg extensions, side planks, the "hundred" exercise, and single-leg bridging. In weeks 4-6, Swiss ball exercises will be introduced, including weight shifting forward and backward, hip flexion, bridging, and contralateral arm.The program will advance in intensity across three phases.
  Arms: Supervised Core Stabilization + Standard Hand Rehabilitation
Behavioral: Unsupervised Core Stabilization + Standard Hand Rehabilitation — he third group will receive the same six-week Standard Hand Rehabilitation Program as the control group (5 days/week for 3 weeks, then 3 days/week for 3 weeks). They will also do an Unsupervised Core Stabilization Exercise Program three times a week for six weeks in the same clinic. Exercises will be the same as the supervised group but done alone using videos without a physiotherapist. The exercises will focus on activating the transversus abdominis and coordinating breathing to improve core stability. Each session includes warm-up, main exercises, and cool-down. In weeks 0-2, exercises include diaphragmatic breathing, transversus activation, curl-ups, and bridging. Weeks 2-4 add cross arm-leg extensions, side planks, the "hundred," and single-leg bridging.Weeks 4-6 introduce Swiss ball exercises, including weight shifting forward and backward, hip flexion, bridging, and contralateral arm lifts. The program will advance in intensity across three phases.
  Arms: Unsupervised Core Stabilization + Standard Hand Rehabilitation

SUMMARY:
Hand injuries carry a high risk due to the constant demands for use and their complex functionality. These injuries often occur as a result of various incidents, including household accidents, occupational hazards, traffic collisions, and sports activities, and they are particularly common among male workers. The severity of hand injuries varies widely, ranging from simple soft tissue damage to serious tendon and nerve lacerations, as well as fractures. The extent of the injury can significantly affect the recovery process and the likelihood of patients regaining their previous functional abilities.There is a strong connection between hand injuries and their impact on both emotional status and functional capacity. Changes in the hand's appearance and restrictions in daily activities can lead to feelings of helplessness, frustration, and psychological stress. In particular, concerns about returning to work can further exacerbate psychological distress in workers. Core stabilization plays a crucial role in alleviating these negative effects. The core region not only ensures overall body stability but also directly influences hand function. Strengthening and stabilizing the core muscles enhance proper body movement, thereby improving upper extremity efficiency. This physical improvement also contributes to psychological recovery, as the ability to perform daily activities more comfortably enhances self-confidence and overall quality of life. Therefore, core exercises do not only improve functional outcomes but also support psychological well-being.

This study will include 51 male patients diagnosed with traumatic hand injuries who meet the inclusion criteria. Assessments will be conducted on joint range of motion, grip strength, joint position sense, reaction time, hand function, activity and participation levels, quality of life, anxiety and depression scales, galvanic skin response, patient satisfaction, and core stability. These evaluations will be performed at two different time points: before rehabilitation and at the end of a six-week rehabilitation program. The study consists of three groups. The first group will participate solely in a standard hand rehabilitation program. The second group will perform supervised core stabilization exercises three times per week in addition to the standard hand rehabilitation program. In the third group, core stabilization exercises will be performed without the supervision of a physiotherapist, with patients following pre-recorded instructional videos alongside the standard rehabilitation program. For all groups, the hand rehabilitation program will take place five days a week for the first three weeks and three days a week for the following three weeks. Patients in the two groups performing core stabilization exercises will be trained in how to activate the transversus abdominis muscle and coordinate their breathing before starting the exercises. The exercises, including warm-up and cool-down phases, will be performed for ten repetitions per session, with each session lasting between 60 and 90 minutes. Additionally, patients will be assigned home exercises from the standard physiotherapy program, and adherence to these exercises will be monitored through checklists.

Although the biomechanical relationship between core muscles and hand function has been explained in the literature, no rehabilitation program incorporating core stabilization exercises for hand injuries has been identified. Moreover, no studies have objectively assessed emotional changes following traumatic hand injuries. This study aims to make a significant contribution to the literature by examining the effects of core stabilization on hand function and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with a traumatic hand injury
* Having received surgical treatment appropriate to the type of injury
* Being a male individual between 20 and 50 years of age
* Having a moderate, severe, or major score according to the Modified Hand Injury Severity Score (MHISS)

Exclusion Criteria:

* Having a chronic illness such as neurological, rheumatological, diabetes, metabolic syndrome, or cardiovascular diseases
* Presence of infection

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Hand Function Assessment (Jebsen-Taylor Hand Function Test) | Before treatment, week 6
Emotional State Assessment (Galvanic Skin Response Device) | Before treatment, week 6
Core Stability Assessment (Stabilizer Biofeedback Device) | Before treatment, week 6

SECONDARY OUTCOMES:
Range of Motion Assessment (Goniometer) | Before treatment, week 6
Proprioception Assessment (Wrist Joint Position Sense Assessment with Goniometer) | Before treatment, week 6
Reaction Time Assessment (Nelson Reaction Time Test) | Before treatment, week 6
Activity and Participation Level Assessment (Disabilities of the Arm, Shoulder and Hand - DASH Questionnaire) | Before treatment, week 6
Severity Evaluation of Hand Injuries (Modified Hand Injury Severity Score) | Baseline (prior to surgery)
Quality of Life Assessment (SF-36) | Before treatment, week 6
Anxiety Assessment (Beck Anxiety Inventory) | Before treatment, week 6
Depression Assessment (Beck Depression Inventory ) | Before treatment, week 6
Patient Satisfaction Assessment (Likert Scale) | Before treatment, week 6
Gross / Fine Grip Strength Assessment (Dynamometer / Pinch meter) | Before treatment, week 6

CONTACTS AND LOCATIONS:
Overall Officials: Gül Deniz YILMAZ YELVAR, Study Chair — Istinye University
Locations (1):
- Istinye University Bahcesehir Liv Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request. Data will be provided for ethically approved, non-commercial research purposes. Interested investigators should contact the principal investigator through the affiliated institution and submit a written request describing the intended use and data handling procedures. Each request will be reviewed individually in accordance with institutional data-sharing guideline.

REFERENCES:
- [Background] Abd-Elfattah HM, Aly SM. Effect of Core Stability Exercises on Hand Functions in Children With Hemiplegic Cerebral Palsy. Ann Rehabil Med. 2021 Feb;45(1):71-78. doi: 10.5535/arm.20124. Epub 2021 Feb 9. PMID 33557483
- [Background] Ayhan C, Unal E, Yakut Y. Core stabilisation reduces compensatory movement patterns in patients with injury to the arm: a randomized controlled trial. Clin Rehabil. 2014 Jan;28(1):36-47. doi: 10.1177/0269215513492443. Epub 2013 Jul 3. PMID 23823711